CLINICAL TRIAL: NCT01062672
Title: Functional Neuroimaging of Cortical Plasticity in the Human Visual System
Status: Withdrawn | Type: Observational
Why Stopped: PI left institution and no participants were enrolled
Sponsor: Baylor College of Medicine (Other)
Collaborators: Brigham and Women's Hospital (Other)
Responsible Party: Principal Investigator, Eli M Mizrahi, Professor, Baylor College of Medicine
Other Study IDs: H--22516
Record Dates: First submitted 2010-02-03; First posted 2010-02-04 (Estimated); Last update posted 2022-04-11 (Actual); Status verified 2022-04

CONDITIONS: Stroke; Blindness; Vision
Keywords: plasticity; reorganization; cortical; fMRI; rehabilitation
MeSH Terms: conditions — Stroke; Blindness

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The study's objective is to measure changes in human visual cortex organization that may arise as a result of injury to the visual pathways. Subjects with retinal or cortical injury will be studied and compared to appropriate controls. Functional magnetic resonance imaging methods are used to monitor cortical topography in time. The main aims of the study are to determine: 1) what are the patterns of cortical reorganization that are seen spontaneously after injury, and 2) whether rehabilitative training can promote adaptive reorganization enhancing recovery.

ELIGIBILITY:
Inclusion Criteria:

* Stable lesion of the visual pathways resulting in a visual field scotoma.

Exclusion Criteria:

* Inability to undergo magnetic resonance imaging,
* Inability to comply with basic instructions,
* Inability to perform the behavioral tasks required,
* Patients with chronic progressive neurological or psychiatric disorders,
* Patients that are pregnant, or breast feeding.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients with lesions of the visual pathway (cortical or retinal)
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2009-01 (Actual); Primary Completion 2015-12 (Actual); Study Completion 2015-12 (Actual)

CONTACTS AND LOCATIONS:
Locations (2):
- Baylor College of Medicine, Houston, Texas, United States
- Max Planck Institute for Biological Cybernetics, Tübingen, Germany